CLINICAL TRIAL: NCT05961683
Title: Evaluating Pressures at the Nares During Non-invasive Ventilation in Newborn Infants Utilizing NIV Plus Software
Brief Title: Evaluating Pressures During Non-invasive Ventilation Utilizing NIV Plus Software
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keck School of Medicine of USC (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Manoj Biniwale, Associate Professor of Pediatrics, Keck School of Medicine of USC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13192
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Distress Syndrome, Newborn; Apnea of Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Infants receiving non invasive ventilation without NIV plus (No Intervention)
- Infants receiving non invasive ventilation with NIV plus (Experimental)
  Interventions: Device: NIV plus software

INTERVENTIONS:
Device: NIV plus software — interventions received by infants studied after placing them on ventilator using NIV plus software
  Arms: Infants receiving non invasive ventilation with NIV plus

SUMMARY:
In the past many neonates with respiratory distress syndrome would require intubation, but over the years these rates have declined as the capabilities of non-invasive ventilation (NIV) have vastly improved. Despite these improvements, the decrease in pressure transmission due to factors such as resistance from tubing or air leaks around the nostrils and mouth, continues to be one of the major drawbacks when using nasal NIV. Current ventilators measure the set pressures at the circuit but do not capture the delivered pressure at the patient's nares. Recently, Medtronic PB980 ventilators feature NIV plus and leak sync software that can be calibrated to measure the pressures provided at the nostrils. Optimum pressures received at the nostrils to provide safe and effective therapy in neonates is currently unknown. In the prospective portion of the study, we aim to evaluate safety and efficacy of the software by comparing the average pressure difference between the circuit and delivery pressure at the nares, the incidence of apnea, bradycardia, desaturations as well as escalation and de-escalation of ventilator support in newborns who are receiving NIV admitted to NICU

ELIGIBILITY:
Inclusion Criteria:

* Gestation Age of 23-41 weeks
* Born at LAC+USC Medical Center and admitted to NICU
* Received NIPPV or nasal CPAP

Exclusion Criteria:

* Infants with any congenital anomalies
* Infants receiving only comfort care measures.
* Infants receiving invasive mode of mechanical ventilation (intubated)
* Non-inborn neonates
* Re-admissions to the NICU

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
interventions performed while using NIV plus software | 24 hours
  will study the number of interventions performed when NIV plus software is used

SECONDARY OUTCOMES:
difference in pressures set and received | 12 hours
  will study the pressure difference as calculated by NIV plus software

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles General Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided